CLINICAL TRIAL: NCT01890785
Title: A Phase 1, Open-label, Randomized, 3-period Crossover Study Evaluating the Relative Bioavailability of SPD489 When the Contents Are Emptied Into a Soft Food and Orange Juice in Healthy Adult Subjects
Brief Title: Bioavailability Study of SPD489 Administered With Two Different Means of Administration in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-123
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lisdexamfetamine Dimesylate Fasting (Experimental): lisdexamfetamine dimesylate 70 mg capsule administered under fasted conditions
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Lisdexamfetamine Dimesylate Vanilla Yogurt (Experimental): Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Lisdexamfetamine Dimesylate Orange Juice (Experimental): Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice
  Interventions: Drug: Lisdexamfetamine Dimesylate

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Single dose of a 70 mg capsule on Day 1
  Other Names: SPD489

SUMMARY:
Compare the pharmacokinetic profiles when the contents are emptied into a soft food and orange juice compared to the SPD489 when swallowed as an intact capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years inclusive at the time of consent. The date of signing informed consent is defined as the beginning of the Screening Period. This inclusion criterion will only be assessed at the first screening visit.
2. Willingness to comply with any applicable contraceptive requirements fo the protocol and is:

   * Male, or
   * Non pregnant, non lactating female
   * Females must be at least 90 days post partum or nulliparous
3. Must be considered "healthy". Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram, hematology, blood chemistry, and urinalysis.
4. An understanding, ability, and willingness to fully comply with study procedures and restrictions
5. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with International Conference on harmonisation Good Clinical Practice Guideline E6 (1996) and applicable regulations, before completing any study related procedures
6. A body mass index between 18.5-30.0kg/m² inclusive. This inclusion criterion will only be assessed at the first screening visit.
7. A hemoglobin value of >=12.0g/dL at the Screening Visit and on Day -1 of Treatment Period 1.
8. Ability to swallow a dose of investigational product according to the study conditions.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria are met at the Screening Visit or at Day 1 of Treatment Period 1 (if reassessed):

1. Current or recurrent disease (eg, cardiovascular, renal, liver, gastrointestinal, malignancy, or other conditions) that could affect the action, absorption, or disposition of the investigational products, or could affect clinical or laboratory assessments.
2. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
3. Significant illness, as judged by the investigator, within 2 weeks of the first dose of investigational product.
4. History of significant anxiety, tension, or agitation as assessed by the investigator.
5. History of or current diagnosis of glaucoma.
6. History of a seizure disorder (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or known family history of Tourette's Disorder.
7. History or presence of known structural cardiac abnormalities, syncope, cardiac conduction problems, exercise-related cardiac events, or clinically significant bradycardia.
8. History of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischemic attack or stroke or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
9. History of controlled or uncontrolled hypertension or a resting supine systolic blood pressure >139mmHg or diastolic blood pressure >89mmHg.
10. Known family history of sudden cardiac death or ventricular arrhythmia.
11. Currently considered a suicide risk, has previously made a suicide attempt, or has a history of, or is currently demonstrating suicidal ideation.
12. Current use of any medication (including prescription, over-the-counter, herbal or homeopathic preparations) with the exception of hormonal replacement therapy or hormonal contraceptives (current use is defined as use within 14 days of first dose of investigational product).
13. Use of any medication known to inhibit or induce the cytochrome P450 (CYP450) enzymes responsible for the metabolism of the investigational product within 14 days of first dose of investigational product.
14. Known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.
15. Known or suspected intolerance or hypersensitivity to orange juice or vanilla yogurt.
16. History of alcohol or other substance abuse within the last year.
17. A positive screen for alcohol or drugs of abuse at the Screening Visit or on Day 1 of Treatment Period 1.
18. Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day. (1 alcohol unit=1 beer=1 wine [5oz]=one liquor [1.5 oz]=0.75oz alcohol.).
19. A positive human immunodeficiency virus antibody screen, Hepatitis B surface antigen, or Hepatitis C virus antibody screen.
20. Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch) within 30 days prior to the first dose of investigational product.
21. Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches or have a history of caffeine withdrawal headaches. (One caffeine unit is contained in the following items: one 6oz cup of coffee, two 12oz cans of cola, one 12oz cup of tea, three 1oz chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine).
22. Donation of blood or blood products (eg, plasma or platelets) within 60 days prior to the first dose of investigational product.
23. Use of another investigational product within 30 days prior to receiving the first dose of investigational product or active enrollment in another drug or vaccine clinical study.
24. Substantial changes in eating habits within 30 days prior to receiving the first dose of investigational product, as assessed by the investigator.
25. An inability to follow a standardized diet and meal schedule or inability to fast, as required during the study.
26. Prior screen failure, randomization, participation, or enrollment in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2013-08-22 (Actual); Study Completion 2013-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Inc, Miami, Florida, United States

REFERENCES:
- [Result] Ermer J, Corcoran M, Lasseter K, Martin PT. Relative Bioavailabilities of Lisdexamfetamine Dimesylate and D-Amphetamine in Healthy Adults in an Open-Label, Randomized, Crossover Study After Mixing Lisdexamfetamine Dimesylate With Food or Drink. Ther Drug Monit. 2016 Dec;38(6):769-776. doi: 10.1097/FTD.0000000000000343. PMID 27661399

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice for first intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt for second intervention; then Lisdexamfetamine Dimesylate 70mg intact capsule fasting for third intervention
- Sequence 2: Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt for first intervention; then Lisdexamfetamine Dimesylate 70mg intact capsule fasting for second intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice for third intervention
- Sequence 3: Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt for first intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice for second intervention; then Lisdexamfetamine Dimesylate 70mg intact capsule fasting for third intervention
- Sequence 4: Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice for first intervention; then Lisdexamfetamine Dimesylate 70mg intact capsule fasting for second intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt for third intervention
- Sequence 5: Lisdexamfetamine Dimesylate 70mg intact capsule fasting for first intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice for second intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt for third intervention
- Sequence 6: Lisdexamfetamine Dimesylate 70mg intact capsule fasting for first intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt for second intervention; then Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice for third intervention
Period: First Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 4 | 5 | 5 | 5 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.6 (10.16) | 35.4 (12.42) | 42.2 (4.44) | 34.2 (12.42) | 39.6 (9.86) | 41.8 (10.06) | 37.6 (10.07)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 65 years, inclusive | 5 | 5 | 5 | 5 | 5 | 5 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 0 | 2 | 2 | 8
  Male | 4 | 3 | 4 | 5 | 3 | 3 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 5 | 5 | 5 | 5 | 5 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) for Lisdexamfetamine Dimesylate
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Up to 96 hours post-dose
Population: Pharmacokinetic Set consisted of all subjects in the Safety Set for whom the primary pharmacokinetic data were considered sufficient and interpretable. Safety Set consisted of subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Groups:
- Lisdexamfetamine Dimesylate Mixed in Orange Juice: Lisdexamfetamine Dimesylate 70mg capsule mixed into orange juice (Single dose of a 70 mg capsule on Day 1)
- Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt: Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt (Single dose of a 70 mg capsule on Day 1)
- Lisdexamfetamine Dimesylate Intact Capsule Fasting: Lisdexamfetamine Dimesylate 70 mg capsule administered under fasted conditions (Single dose of a 70 mg capsule on Day 1)
Arm/Group | Lisdexamfetamine Dimesylate Mixed in Orange Juice | Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt | Lisdexamfetamine Dimesylate Intact Capsule Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng*hr/ml | 27.0 (7.8) | 36.0 (14.2) | 38.3 (12.3)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate Mixed in Orange Juice vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.708, 90% CI 2-sided [0.655 to 0.766]
Statistical Analysis 2: Comparison: Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.918, 90% CI 2-sided [0.849 to 0.992]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for Lisdexamfetamine Dimesylate
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Up to 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lisdexamfetamine Dimesylate Mixed in Orange Juice | Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt | Lisdexamfetamine Dimesylate Intact Capsule Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng/ml | 24.5 (7.48) | 32.2 (11.46) | 38.5 (13.07)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate Mixed in Orange Juice vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.641, 90% CI 2-sided [0.582 to 0.707]
Statistical Analysis 2: Comparison: Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.828, 90% CI 2-sided [0.752 to 0.912]

3. Primary Outcome: AUC for D-amphetamine
Description: d-Amphetamine is a metabolite of Lisdexamfetamine Dimesylate and is an active form that is responsible for the drug's therapeutic activity.
Time Frame: Up to 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Lisdexamfetamine Dimesylate Mixed in Orange Juice | Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt | Lisdexamfetamine Dimesylate Intact Capsule Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng*h/ml | 1140.9 (274.1) | 1110.1 (252.9) | 1180.2 (295.1)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate Mixed in Orange Juice vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.970, 90% CI 2-sided [0.937 to 1.004]
Statistical Analysis 2: Comparison: Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.944, 90% CI 2-sided [0.912 to 0.977]

4. Primary Outcome: Cmax for D-amphetamine
Description: as for outcome 3
Time Frame: Up to 96 hours-post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lisdexamfetamine Dimesylate Mixed in Orange Juice | Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt | Lisdexamfetamine Dimesylate Intact Capsule Fasting
Number analyzed (Participants) | 30 | 30 | 30
ng/ml | 59.1 (9.47) | 59.0 (9.28) | 61.0 (10.81)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate Mixed in Orange Juice vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.971, 90% CI 2-sided [0.945 to 0.998]
Statistical Analysis 2: Comparison: Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt vs Lisdexamfetamine Dimesylate Intact Capsule Fasting; Test type: Superiority or Other; Ratio of geometric least squares means = 0.970, 90% CI 2-sided [0.944 to 0.997]

ADVERSE EVENTS:
Groups:
- Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt: Lisdexamfetamine Dimesylate 70mg capsule mixed into vanilla yogurt(Single dose of a 70 mg capsule on Day 1)
Arm/Group | Lisdexamfetamine Dimesylate Mixed in Orange Juice | Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt | Lisdexamfetamine Dimesylate Intact Capsule Fasting
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 16/30 | 17/30 | 9/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate Mixed in Orange Juice (N=30) | Lisdexamfetamine Dimesylate Mixed in Vanilla Yogurt (N=30) | Lisdexamfetamine Dimesylate Intact Capsule Fasting (N=30)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 5 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 8 (8) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 4 (4)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.